CLINICAL TRIAL: NCT04992156
Title: A Retrospective Study of Prediction of 18F-FES-PET/CT Parameters on the Outcome of Palbociclib Combined With Endocrine Therapy in Patients With HR+ and HER2-metastatic Breast Cancer
Brief Title: Prediction of 18F-FES-PET/CT Parameters on Palbociclib Combined With ET
Status: Completed | Type: Observational
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Biyun Wang, MD, Professor, Fudan University
Other Study IDs: YOUNGBC-15
Record Dates: First submitted 2021-08-01; First posted 2021-08-05 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients cohort: Patients with MBC in the Fudan University Shanghai Cancer Center who underwent whole-body 18F-FES PET/CT before the initiation of Palbociclib was included.
  Interventions: Drug: Palbociclib

INTERVENTIONS:
Drug: Palbociclib — Palbociclib 125mg/d

SUMMARY:
To investigate parameters based on 18F-FES-PET/CT so as to estimate the outcome of palbociclib combined with endocrine therapy in patients with HR+/HER2-MBC.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients aged 18-70 years.
2. Metastatic breast cancer included unresectable locally advanced breast cancer, de novo stage IV breast cancer, and recurrent metastatic breast cancer.
3. HR+ was defined as estrogen receptor- or progesterone receptor-positive status by immunohistochemistry.
4. HER2 status was determined by immunohistochemistry or fluorescence in situ hybridization.
5. Palbociclib treatment of metastatic breast cancer for at least one cycle.
6. Available medical history.

Exclusion Criteria:

1.Incomplete medical history.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with breast cancer with confirmed metastasis, regardless of being de novo diagnosed or progressed from a non-metastatic stage.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2017-03-15 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-04-15 (Actual)

PRIMARY OUTCOMES:
PFS | Through study completion, an expected average of 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Biyun Wang, Dr, Principal Investigator — Fudan University
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

REFERENCES:
- [Derived] Liu C, Hu S, Xu X, Zhang Y, Wang B, Song S, Yang Z. Evaluation of tumour heterogeneity by 18F-fluoroestradiol PET as a predictive measure in breast cancer patients receiving palbociclib combined with endocrine treatment. Breast Cancer Res. 2022 Aug 26;24(1):57. doi: 10.1186/s13058-022-01555-7. PMID 36028895